CLINICAL TRIAL: NCT03915691
Title: Isthmus Guided vs Anatomical Linear Ablation in the Treatment of Scar Related Atrial Tachycardia
Brief Title: The RIPPLE AT-PLUS Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Norfolk & Norwich University Hospital Trust (Unknown); Nottingham University Hospitals NHS Trust (Other); University Hospitals Plymouth NHS Trust (Unknown); Blackpool Teaching Hospitals NHS Trust (Unknown); Cardiff & Vale UHB (Unknown); University Hospitals Sussex NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19SM5013
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Atrial Tachycardia
Keywords: Atrial Tachycardia; Atrial Fibrillation; Mapping; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isthmus targeted approach using Ripple Mapping (Active Comparator): Intervention: Isthmus targeted approach using Ripple Mapping catheter ablation of atrial tachycardia.
  Interventions: Procedure: Catheter ablation of atrial tachycardia: Ripple Mapping guided.
- Conventional Mapping (Active Comparator): Intervention: conventional catheter ablation of atrial tachycardia.
  Interventions: Procedure: Catheter ablation of atrial tachycardia: Conventional mapping guided.

INTERVENTIONS:
Procedure: Catheter ablation of atrial tachycardia: Ripple Mapping guided. — Ripple Mapping is used to map the atrial tachycardia mechanism. Using the scar thresholding technique the Ripple Map is interpreted and catheter ablation directed to the site of the heart identified as putative to the arrhythmia mechanism. All ablation lesions are confirmed to have conduction block across them using Ripple Mapping. This can include lesions created at previous ablation procedures.
  Arms: Isthmus targeted approach using Ripple Mapping
Procedure: Catheter ablation of atrial tachycardia: Conventional mapping guided. — Conventional activation mapping is used to map the atrial tachycardia mechanism. The resultant (activation) map is interpreted and ablation directed to the site of the heart identified as putative to the arrhythmia mechanism. All ablation lesions are confirmed to have conduction block across them using conventional mapping. This can include lesions created at previous ablation procedures.
  Arms: Conventional Mapping

SUMMARY:
Atrial tachycardia is a symptomatic arrhythmia, for which an effective treatment is a catheter ablation procedure. The goal of the Ripple AT-Plus study is to evaluate two methods of performing catheter ablation for atrial tachycardia. The main outcome assessed during the study is long-term recurrence of atrial tachycardia following the catheter ablation procedure.

DETAILED DESCRIPTION:
Catheter based mapping of the electrical signals in the heart during atrial tachycardia can identify areas that require ablation in order to treat the arrhythmia. There are numerous methods by which to map atrial tachycardia. Isthmus guided ablation using Ripple Mapping is one such method, and has recently been demonstrated to improve diagnostic accuracy of mapping and therefore improve acute procedural outcomes (termination of the tachycardia).

However, it is not known if improved acute procedural outcomes translate into long-term benefits for patients. At present, the recurrence rate following atrial tachycardia ablation is near 30%. We hypothesise that isthmus guided ablation using Ripple Mapping can reduce long-term recurrence following ablation as improved diagnostic accuracy of mapping can lead to more targeted, less extensive, ablation.

Patients referred for catheter ablation of atrial tachycardia will be randomised to undergo the procedure by isthmus targeted approach using Ripple Mapping or conventional approach using local activation time. Otherwise, the catheters used to perform the mapping and ablation will be the same in both groups. After the procedure, follow up will occur at 1 year with a further Holter Montior. Any arrhythmia recurrence will be documented and the two arms will be compared for acute success, 12 month success, ablation required and procedure time.

ELIGIBILITY:
Inclusion Criteria:

1. Referred for catheter ablation of AT by the direct care team, based on clinical indication.
2. Male or female, aged >18 years old.
3. Able to consent for recruitment to the trial and the catheter ablation procedure.

Exclusion Criteria:

1. Contraindication to catheter ablation as deemed by the clinical team.
2. Typical atrial flutter or AF on ECG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Atrial arrhythmia recurrence | 12 months
  Any confirmed episode of atrial arrhythmia (>30 seconds on Holter or 12 lead ECG) occurring in the 12 months after catheter ablation.

SECONDARY OUTCOMES:
Acute success during the catheter ablation procedure by the first ablation set. | Procedure.
  Atrial tachycardia termination (acute success) during ablation delivered to only target the diagnosed AT mechanism by the mapping approach used (first ablation set).
Acute success during the catheter ablation procedure without the need of entrainment. | Procedure.
  Entrainment not required to confirm or exclude the diagnosis made by 3D electroanatomic mapping methods.
Procedure failure. | Procedure.
  Inability to terminate atrial tachycardia during the catheter ablation procedure, requiring external electrical cardioversion to achieve sinus rhythm.
Total procedure time. | Procedure.
  Procedure time measured from initiation of intracardiac mapping to catheter removal from the body.
Ablation required | Procedure.
  Ablation required, measured using pre-defined ablation index or ablation line length.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Luther, MBBS, Principal Investigator — Liverpool Heart & Chest Hospital
Locations (3):
- United Kingdom (3):
  - Liverpool Heart & Chest Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Freeman Hospital, The Newcastle Upon Tyne NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kailey B, Kemp I, Taylor M, Crooks J, Katritsis G, Koa-Wing M, Jamil-Copley S, Linton N, Kanagaratnam P, Gupta D, Luther V. Ripple AT Plus - isthmus-guided vs conventional ablation in the treatment of scar-related atrial tachycardia: study protocol for a randomised controlled trial. J Interv Card Electrophysiol. 2023 Oct;66(7):1533-1539. doi: 10.1007/s10840-023-01607-8. Epub 2023 Aug 18. PMID 37594646